CLINICAL TRIAL: NCT05574361
Title: A Prospective Multi-Center Continued Access Protocol for the Use of the LifePort® Liver Transporter (LLT) System With Vasosol® in Orthotopic Liver Transplants (PILOT™_CA: Perfusion to Improve Liver Outcomes in Transplantation_ Continued Access Arm)
Brief Title: Continued Access Study to Evaluate Performance of the Organ Recovery Systems _LifePort® Liver Transporter System, a Machine Perfusion System, for Liver Transplant (PILOT™_CA)
Acronym: PILOT™_CA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Organ Recovery Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-US-02-ORS
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Hypothermic Machine Perfusion (Experimental): Hypothermic Machine Perfusion with Organ Recovery Systems LifePort Liver Transporter system
  Interventions: Device: Hypothermic Machine Perfusion

INTERVENTIONS:
Device: Hypothermic Machine Perfusion — Organ Recovery Systems LifePort® Liver Transporter (LLT) System and Vasosol® Machine Perfusion Solution

SUMMARY:
To provide continued access for the LLT system to provide additional safety data in support of the PILOT pivotal efficacy and safety trial

DETAILED DESCRIPTION:
To provide continued access for the LLT System with Vasosol® for the preservation of whole explanted livers, thereby providing additional safety data in support of the PILOT pivotal efficacy and safety trial

ELIGIBILITY:
* ≥18 years of age.
* Active on the United Network for Organ Sharing (UNOS) waiting list for liver transplantation.
* De novo liver transplant recipient.
* Written informed consent required.

Exclusion Criteria:

* Subject is a multi-organ transplant recipient.
* Subject is antibodies blood group (ABO) liver incompatible.
* Subject has severe systemic infection.
* Subject is Human Immunodeficiency Virus (HIV) positive.
* Subject has acute/fulminant liver failure.
* Subject is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Early Allograft Dysfunction (EAD) | 7 days
  EAD defined as total bilirubin ≥ 10 mg/dL or International Normalized Ratio (INR) ≥ 1.6 or Aspartate Aminotransferase (AST) >2000IU/L or Alanine Aminotransferase (ALT) > 2000 IU/L

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Lindower, Study Director — Organ Recovery Systems; Matthew Copithorne, Study Chair — Organ Recovery Systems
Locations (5):
- United States (5):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Intermountain Medical Center, Murray, Utah

IPD SHARING:
Plan to Share IPD: No